CLINICAL TRIAL: NCT06272149
Title: An Exploratory Clinical Trial to Evaluate the Tolerability and Safety of VGN-R08b Via Intracerebroventricular Injection in Patients With Type II Gaucher Disease
Brief Title: An Exploratory Clinical Trial of VGN-R08b in Patients With Type II Gaucher Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGN-R08b-001
Record Dates: First submitted 2023-07-17; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-02

CONDITIONS: Type II Gaucher Disease
Keywords: GBA, Glucocerceramide, AAV9, CNS gene therapy
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- type II Gaucher disease (Experimental): This is a single-center, open, dose-climbing investigator-sponsored exploratory clinical study that included a dose-climbing phase and a dose-expanding phase. The sponsor plans to explore two dose levels in dose-climbing phase (one subject each cohort), then have additional 2~4 subjects in dose-expanding phase
  Interventions: Drug: VGN-R08b

INTERVENTIONS:
Drug: VGN-R08b — VGN-R08b is a kind of Gene therapy with adeno-associated virus (AAV) serotype 9 (AAV9) driven human GBA1 being injected directly into intracerebroventricular.

SUMMARY:
This exploratory trial is to prove the tolerability and safety of VGN-R08b to treat infants with type II Gaucher disease.

DETAILED DESCRIPTION:
Gaucher disease (GD) is an autosomal recessive genetic metabolic disorder. Due to the mutation of Glucocerebrosidase gene (GBA1), the activity of glucocerebrosidase (GCase) in the lysosome of the body is reduced, causing its substrate glucocerceramide to be accumulated in macrophage lysosomes in the liver, spleen, bone, lung, brain and eyes. Type II, acute neuropathy, with extensive and severe visceral involvement, usually develops within the first year of life, and most children die before the age of 2. VGN-R08b is a kind of Gene therapy with adeno-associated virus (AAV) serotype 9 (AAV9) driven human GBA1 being injected directly into intracerebroventricular.

This is a single-center, open, dose-climbing investigator-sponsored exploratory clinical study that included a dose-climbing phase and a dose-expanding phase. The sponsor plans to explore two dose levels in dose-climbing phase (one subject each cohort), then have additional 2~4 subjects in dose-expanding phase.

This study is to give preliminary evidence for the safety and efficacy of VGN-R08b treatment for patients with type II Gaucher disease.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with age of ≤24 months.
2. Historical diagnosis of Gaucher disease confirmed by GCase enzyme activity test, and with GBA1 biallelic mutations.
3. Neurological signs and/or symptoms consistent with diagnosis of GD2.
4. Parent(s)/legal guardian(s) of subject must give their consent for subject to enroll in the study.
5. Parent(s)/legal guardian(s) of the subject must agree to comply with the requirements of the study, including providing disease information and support disease assessment of symptoms.

Exclusion Criteria:

1. Diagnosis of a significant CNS disease other than GD2 that may be a cause for the patient's GD symptoms or may confound study objectives.
2. Achieved independent gait.
3. Severe visceral symptoms of GD which, in the opinion of the Investigator, would pose an unacceptable risk to the patient or interfere with the patient's ability to comply with study procedures or interfere with the conduct of the study.
4. Clinically active infection (including HIV, HBV, HCV or syphilis).
5. For those receiving enzyme replacement therapy and/or substrate reduction therapy and/or ambroxol for Gaucher disease, stable treatment ≤2 months before enrollment.
6. Use of strong inhibitors or inducers of cytochrome CYP3A4 or P-glycoprotein (P-gp) medications, herbals, or over-the-counter agents.
7. Any type of prior gene or cell therapy.
8. Immunizations (live vaccines) in the prior 4 weeks.
9. Use of systemic immunosuppressant or corticosteroid therapy other than protocol-specified (topical preparations for dermatological conditions are allowed).
10. Patients with anti-AAV9 neutralizing antibody titer over 1:5.
11. Brain MRI (magnetic resonance imaging) showing clinically significant abnormality considered to prevent intracisternal injection.
12. Contraindication to sedation during surgery or imaging studies (PET).
13. Presence of other significant medical conditions that would create an unacceptable risk to the patient or interfere with the patient's ability to comply with study procedures or interfere with the conduct of the study.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) | Week 52
  Adverse Events (AEs), Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Long-term safety follow-up | Up to Year 5
  Number of Adverse Events (AEs), Serious Adverse Events (SAEs)
Survival ratio at age of 24 months | Baseline until event, or reach the age of 24 months, Up to Year 5
  Survival ratio at age of 24 months
Changes in the activity of glucose cerebroside lipase (GCase) | Up to Year 5
  Pharmacodynamic indicators
Changes in the activity of glucose cerebroside (GC) levels | Up to Year 5
  Pharmacodynamic indicators
Changes in the activity of glucose sphingosine (Lyso GL1) levels in peripheral blood and CSF after medication | Up to Year 5
  Pharmacodynamic indicators
Immunogenicity | 26 weeks
  Number of subjects producing antibodies against AAV9 and GCase
Changes in the genomic level of VGN-R08b vector in peripheral blood after medication | 26 weeks
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Huiwen, Dr., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No